CLINICAL TRIAL: NCT02309203
Title: Canadian Study of the MicroVention Flow Re-Direction (FRED) Endoluminal Device Stent System in the Treatment of Intracranial Aneurysms - The CanFRED Trial
Brief Title: Canadian Study of the MicroVention Flow Re-Direction (FRED) Endoluminal Device Stent System in the Treatment of Intracranial Aneurysms
Acronym: CanFRED
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not initiated at our site.
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Principal Investigator, Jean Raymond, MD, Centre hospitalier de l'Université de Montréal (CHUM)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE 14.295
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Intracranial Aneurysms
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Flow Re-Direction Endoluminal Device (Experimental): Flow Re-Direction Endoluminal Device (FRED Device)
  Interventions: Device: FRED

INTERVENTIONS:
Device: FRED — Flow Re-Direction Endoluminal Device

SUMMARY:
The study objective is to evaluate the safety and effectiveness of the MicroVention FRED System when used in the treatment of wide-necked intracranial aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* Subject whose age is ≥ 18 years;
* Subject has a single target aneurysm located in the following zones:
* Zone 1 - Petrous through cavernous of the ICA
* Zone 2 - Ophthalmic segment of the ICA
* Zone 3-Posterior Circulation, basilar artery (not including the basilar bifurcation), vertebral artery
* Subjects with a single target intracranial aneurysm located along the internal carotid artery, or the vertebral or basilar artery for whom existing endovascular options (coiling, stent-assisted-coiling) could be ineffective or because aneurysm is predisposed to recurrence due to having any of the following characteristics:
* Aneurysms with a neck > 4mm, dome to neck ratio ≤2 or no discernible neck
* Fusiform aneurysms of any size requiring treatment;
* The parent artery must have a diameter of 2.5 - 5.0mm distal/proximal to the target intracranial aneurysm (IA);
* Subject fulfills study requirements, and the subject or his/her legally authorized representative provides a signed informed consent form;
* Negative pregnancy test in a female subject who has had menses in the last 24 months;
* Subject is willing to return for the 1-month and 6-month follow-up evaluations

Exclusion Criteria:

* Subject who is pregnant or breastfeeding; Subject who suffers from a subarachnoid hemorrhage in the last 60 days;
* Subject who suffers from any intracranial hemorrhage in the last 30 days;
* Subject currently undergoing radiation therapy for carcinoma or sarcoma of the head or neck region;
* Subject with stenosis of the parent artery (>50%) proximal to the target aneurysm;
* Subject with known platelet dysfunction or a contraindication to or inability to tolerate anticoagulants/antiplatelet agents;
* Subject with contraindications or severe allergies to anticoagulants or antiplatelet medications (aspirin, heparin, ticlopidine, clopidogrel, prasugrel or ticagrelor);
* Subject with known hypersensitivity to metal, such as nickel-titanium and metal jewelry
* Subject with documented contrast allergy, or other condition, that prohibits imaging.
* Evidence of active bacterial infection at the time of treatment;
* Subject who has had a previous intracranial stenting procedure associated with the target aneurysm;
* Subject with life-threatening diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2017-02 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
death or major stroke | within 30 days post procedure
  A major stroke is defined as a new neurological event that persists for > 24 hours and results in a mRS >2. A minor stroke is defined as a new neurological event that persists for > 24 hours.
neurological death or major ipsilateral stroke, measured by mRS. | within 6 months post procedure

SECONDARY OUTCOMES:
Incidence of FRED System and procedure related Serious Adverse Events; | 1 year
Incidence of successful delivery of the FRED System implant; | 24 hours
Incidence of migration of the FRED System implant | 6 months
Unplanned alternative treatment on the target IA (Defined as re-treatment of the target aneurysm due to worsening of the clinical condition of the subject) | Within 6 months
  Defined as re-treatment of the target aneurysm due to worsening of the clinical condition of the subject
Change in clinical and functional outcomes (as measured by an increase in the modified Rankin Scale compared to baseline) | 6 months
  as measured by an increase in the modified Rankin Scale compared to baseline